CLINICAL TRIAL: NCT06750861
Title: QL1706 in Combination With Nab-paclitaxel and Gemcitabine as First-line Treatment in Patients With Locally Advanced or Metastatic Pancreatic Ductal Adenocarcinoma : A Single-arm, Phase II Study
Brief Title: QL1706 Plus Chemotherapy With AG Regime as First-line Treatment of Advanced PDAC
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, LIN YANG, Prof, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC5035
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Pancreatic Adenocarcinoma
Keywords: QL1706; Efficacy; Pancreatic cancer; Safety; Chemotherapy; First-Line
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- QL1706+AG (Experimental): QL1706+AG
  Every 3 weeks as a cycle:
  QL1706: 5mg/kg, IV, D3; Q3W Nab-paclitaxel: 125mg/m2, IV，D1、8; Q3W Gemcitabine: 1000mg/m2，IV，D1、8; Q3W Re-evaluate patients every two cycles. If the patient has been treated for more than 8 cycles, they will enter maintenance therapy, and the regimen is QL1706 monotherapy.
  Interventions: Drug: QL1706

INTERVENTIONS:
Drug: QL1706 — QL1706+AG

SUMMARY:
This is a single-center, open-label, exploratory study to evaluate the efficacy and safety of QL1706 plus nab-paclitaxel and gemcitabine as first-line treatment in patients with unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma.

DETAILED DESCRIPTION:
This study is an open, single-center, exploratory clinical trial designed to evaluate the efficacy and safety of QL1706 in combination with nab-paclitaxel and gemcitabine for the first-line treatment of patients with unresectable locally advanced or metastatic pancreatic ductal adenocarcinoma, who had not received prior systemic therapy.

Subjects sign informed consent, undergo a screening period of examination and evaluation, which lasts for 21 days, and those who meet the entry criteria enter the treatment period and receive QL1706 in combination with albumin-paclitaxel and gemcitabine in 3-week intervals until protocol-specified treatment termination Event. Subjects will be enrolled in the study and wil undergo safety visit prior to D1 dosing for each treatment cycle. lmaging exams and assessments will be performed every 6 weeks (± 7 days) until disease progression, initiation of new anti-tumor therapy, withdrawal of informed consent, or death, whichever occurs first, as confirmed per REClST v1.1. Additional imaging and evaluation may be performed at any time during the study if clinically indicated.

Subjects wil be required to complete safety examinations and imaging assessments at the end of treatment, followed by a safety visit and follow-up until 90 days after the last dose of QL1706 or 30 days after the last dose of other investigational agents, whichever is longer. Survival follow-up is performed after the safety visit, every 60 days (±7 days), to collect and record the subject's survival status and subsequent anti-tumor therapy.The study used ORR as the primary endpoint and was planned to enroll 30 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18, male or female;
2. Has histologically or cytologically confirmed pancreatic ductal adenocarcinoma (PDAC);
3. Has not received prior systemic treatment for their locally advanced or metastatic PDAC;
4. Has presence of measurable disease as defined by Response Evaluation Criteria in Solid Tumours (RECIST 1.1);
5. Has a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Status;
6. Has a life expectancy of at least 3 months;
7. Has adequate organ function;
8. If female of childbearing potential, have a negative serum pregnancy test within 7 days prior to first trial treatment;
9. If female of childbearing potential or a male subject with a partner with childbearing potential, be willing to use a highly effective method of contraception (with a failure rate of less than 1.0% per year) from first study treatment to 24 weeks after completion of the trial treatment.

Exclusion Criteria:

1. Untreated active CNS metastasis or leptomeningeal metastasis.
2. Is currently participating and receiving an investigational drug or has participated in a study of an investigational drug within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first dose of trial treatment;
3. Has received other anti-tumor treatment within 4 weeks or within 5 times of half-life (no less than 2 weeks), whichever is shorter prior to the first trial treatment;
4. Major surgery for any reason, except diagnostic biopsy, within 4 weeks of the first administration of trial treatment and/or if the subject has not fully recovered from the surgery within 4 weeks of the first administration of trial treatment;
5. Curative radiation within 3 months of the first dose of trial treatment. Radiation to more than 30% of the bone marrow or with a wide field of radiation should not be used within 4 weeks prior to the first administration of trial treatment;
6. Subjects receiving immunosuppressive agents (such as steroids) for any reason should be tapered off these drugs before initiation of trial treatment (with the exception of subjects with adrenal insufficiency, who may continue corticosteroids at physiologic replacement doses, equivalent to < 10 mg prednisone daily, inhaled steroids and topical use of steroids);
7. Vaccination within 28 days of the first administration of trial treatment, except for administration of inactivated vaccines (e.g., inactivated influenza vaccines);
8. Has interstitial lung disease, or a history of pneumonitis that required oral or intravenous glucocorticoids to assist with management;
9. History or current active autoimmune disease that might deteriorate when receiving an immunostimulatory agent；
10. Previous malignant disease History of uncontrolled intercurrent illness Prior therapy with any antibody/drug targeting T cell coregulatory proteins Known severe hypersensitivity reactions to antibody drug；
11. Is pregnant or breastfeeding;
12. Other medical conditions that at the discretion of investigator interfere with the requirements of the trial in terms of safety or efficacy evaluation, or treatment compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-15 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 1 year
  ORR of regimen of QL1706+AG
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 1 year
  The incidence and severity (graded by CTCAE 5.0) of treatment emergent adverse events (TEAEs) and treatment-related adverse events (TRAEs), immune-related adverse events ( irAEs).

SECONDARY OUTCOMES:
Median Progression-Free Survival (mPFS) | 1 year
Median Overall Survival (mOS) | 2 years
Duration of Response (DoR) | 1 year
Disease Control Rate (DCR) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, Chaoyang District, China

IPD SHARING:
Plan to Share IPD: No